CLINICAL TRIAL: NCT01491737
Title: A Randomized, Two-Arm, Open-Label, Multicenter Phase II Trial Assessing the Efficacy and Safety of Pertuzumab Given in Combination With Trastuzumab Plus an Aromatase Inhibitor in First Line Patients With HER2-Positive and Hormone Receptor-Positive Advanced (Metastatic or Locally Advanced) Breast Cancer
Brief Title: A Study of Pertuzumab in Combination With Trastuzumab Plus an Aromatase Inhibitor in Participants With Metastatic Human Epidermal Growth Factor Receptor 2 (HER2)-Positive and Hormone Receptor-Positive Advanced Breast Cancer
Acronym: PERTAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO27775; 2011-002132-10 (EudraCT Number)
Record Dates: First submitted 2011-12-06; First posted 2011-12-14 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab; Aromatase Inhibitors; Induction Chemotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy (Experimental): Participants will receive pertuzumab in combination with trastuzumab plus aromatase inhibitor (AI) until pre-defined study end, disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Participants may also receive induction chemotherapy (docetaxel every 3 weeks or paclitaxel weekly) up to the first 18-24 weeks of the treatment period at the investigator's discretion.
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Aromatase Inhibitor; Drug: Induction Chemotherapy
- Arm B: Trastuzumab + AI +/- Chemotherapy (Active Comparator): Participants will receive trastuzumab plus aromatase inhibitor (AI) until predefined study end, disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Participants may also receive induction chemotherapy (docetaxel every 3 weeks or paclitaxel weekly) up to the first 18-24 weeks of the treatment period at the investigator's discretion.
  Interventions: Drug: Trastuzumab; Drug: Aromatase Inhibitor; Drug: Induction Chemotherapy

INTERVENTIONS:
Drug: Pertuzumab — Participants will receive a loading dose of 840 milligrams (mg) as an intravenous infusion on Day 1 of first treatment cycle, followed by 420 mg on Day 1 or Day 2 of each subsequent 3-week cycle until disease progression or unacceptable toxicity.
  Other Names: Perjeta®; rhuMAb 2C4
  Arms: Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy
Drug: Trastuzumab — Participants will receive a loading dose of 8 milligrams per kilogram (mg/kg) as an intravenous infusion on Day 1 or 2 of first treatment cycle, followed by 6 mg/kg on Day 1 or Day 2 of each subsequent treatment 3-week cycles until disease progression or unacceptable toxicity.
  Other Names: Herceptin®; rhuMAb HER2
Drug: Aromatase Inhibitor — Participants will receive 1 mg anastrozole or 2.5 mg letrozole orally once daily.
Drug: Induction Chemotherapy — Participants receiving induction chemotherapy up to the first 18-24 weeks of the treatment period will receive a taxane (docetaxel every 3 weeks or paclitaxel weekly), administered in line with the respective pertuzumab and/or trastuzumab infusions at the investigator's discretion.

SUMMARY:
This randomized, open-label, two-arm, multi-center, Phase II study will evaluate the efficacy and safety of pertuzumab in combination with trastuzumab plus an aromatase inhibitor (AI) in first-line participants with HER2-positive and hormone receptor-positive advanced breast cancer. Participants will be randomized to one of two treatment arms; Arm A (pertuzumab in combination with trastuzumab plus an AI) or Arm B (trastuzumab plus an AI). Participants may also receive induction chemotherapy (a taxane, either docetaxel or paclitaxel) at the investigator's discretion in combination with the assigned treatment arm. The anticipated time on study treatment is until disease progression, unacceptable toxicity, withdrawal of consent, or death whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Participants with HER2-positive and hormone receptor-positive advanced metastatic or locally advanced breast cancer
* Post-menopausal status over 1 year
* HER2-positive as assessed by local laboratory on primary or metastatic tumor
* Hormone-receptor positive defined as estrogen receptor-positive and/or progesterone receptor-positive
* At least one measurable lesion and/or non-measurable disease evaluable according to Response Evaluation Criteria In Solid Tumors Version 1.1

Exclusion Criteria:

* Previous systemic non-hormonal anticancer therapy in the metastatic or locally advanced breast cancer setting
* Previous treatment with anti-HER2 agents for breast cancer, except trastuzumab and/or lapatinib in the neoadjuvant or adjuvant setting
* Disease progression while receiving adjuvant trastuzumab and/or lapatinib treatment
* History of persistent Grade 2 or higher hematological toxicity according to National Cancer Institute-Common Toxicity Criteria Version 4.0
* Disease-free interval from completion of adjuvant/neo-adjuvant systemic non-hormonal treatment to recurrence of within 6 months
* Other malignancies within the last 5 years, except for carcinoma in situ of the cervix or basal cell carcinoma
* Clinical or radiographic evidence of central nervous system metastases or significant cardiovascular disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2012-02-17 (Actual); Primary Completion 2016-03-17 (Actual); Study Completion 2019-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (82):
- United States (21):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Ironwood Cancer TX & Rsch Ctrs, Chandler, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Comprehensive Blood & CA Ctr; Research, Bakersfield, California
  - Rocky Mountain Cancer Center - Denver, Denver, Colorado
  - Norwalk Hospital, Norwalk, Connecticut
  - Advanced Medical Specialties, Miami, Florida
  - Georgia Cancer Specialists - Northside, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, a Service of WellStar Cobb Hospital, Marietta, Georgia
  - Cancer Center of Kansas, Wichita, Kansas
  - Crescent City Rsrch Cnsrtm, LLC, Marrero, Louisiana
  - Weinberg CA Inst Franklin Sq, Baltimore, Maryland
  - Center For Cancer and Blood Disorders, Bethesda, Maryland
  - Washington University School of Medicine; Internal Medicine - Renal, St Louis, Missouri
  - Hematology Oncology Associates; Carol G. Simon Ctr, Morristown, New Jersey
  - Cooper Hospital; Hematology & Oncology, Voorhees Township, New Jersey
  - NS-Long Island Jewish Hlth Sys, Lake Success, New York
  - ProHEALTH Care Associates LLP, Lake Success, New York
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Baylor College of Medicine; Lester & Sue Smith Breast Ctr, Houston, Texas
  - Scott and White Hospital; Cancer Center, Temple, Texas
- Brazil (4):
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Perola Byington, São Paulo, São Paulo
  - Inst. Brasileiro de Controle Ao Cancer; Oncologia Clinica / Quimioterapia, São Paulo, São Paulo
  - Hospital Sao Jose, São Paulo, São Paulo
- France (10):
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Clinique Tivoli; Sce Radiotherapie, Bordeaux
  - Hopital Morvan; Oncologie - Radiotherapie, Brest
  - Centre Jean Perrin; Oncologie, Clermont-Ferrand
  - Clinique De La Sauvegarde; Chimiotherapie, Lyon
  - Centre Catherine de Sienne; Chimiotherapie, Nantes
  - Centre Antoine Lacassagne; Hopital De Jour A2, Nice
  - CH De Senlis; Medecine 2, Senlis
  - Clinique Pasteur; Oncologie Medicale, Toulouse
  - Centre Alexis Vautrin; Oncologie Medicale, Vandœuvre-lès-Nancy
- India (5):
  - Bangalore Institute of Oncology, Bangalore, Karnataka
  - Jaslok Hospital & Research Centre; Medical Oncology, Mumbai, Maharashtra
  - Indraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
  - Apollo Speciality Hospital, Chennai
  - Ruby Hall Clinic, Pune
- Italy (15):
  - Irccs Ist. Tumori Giovanni Paolo Ii; Dipartimento Oncologia Medica, Bari, Apulia
  - Ospedale Antonio Perrino; Oncologia Medica, Brindisi, Apulia
  - Ospedale Vito Fazzi; Div. Oncoematologia, Lecce, Apulia
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Università degli Studi Federico II; Clinica di Oncologia Medica, Napoli, Campania
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi; Unità Operativa Oncologia Medica, Bologna, Emilia-Romagna
  - Ospedale Regionale Di Parma; Divisione Di Oncologia Medica, Parma, Emilia-Romagna
  - A.O. Santa Maria Degli Angeli; U.O Di Oncologia Medica, Pordenone, Friuli Venezia Giulia
  - Ospedale S.S. Trinità Nuovo; Divisione Oncologia, Sora, Lazio
  - Casa di Cura MultiMedica Ospedale di Castellanza; UO Senologia Medica, Castellanza, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 1, Milan, Lombardy
  - IRCCS Fondazione Maugeri; Oncologia Medica I, Pavia, Lombardy
  - Az Ospedaliera Nuovo Garibaldi Quartiere Nesima; Oncologia Medica, Catania, Sicily
  - A.O. Careggi; Radioterapia, Florence, Tuscany
  - Ospedale Misericordia E Dolce; Oncologia Medica, Prato, Tuscany
- Spain (16):
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Hospital Provincial de Castellon; Servicio de Oncologia, Castellon, Castellon
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - IInstituto Oncologico de San Sebastian, Oncologikoa; Servicio de Oncologia, Donostia / San Sebastian, Guipuzcoa
  - Hospital de Donostia; Servicio de Oncologia Medica, Donostia / San Sebastian, Guipuzcoa
  - Complejo Hospitalario Universitario A Coruña (CHUAC, Materno Infantil), Oncología, A Coruña
  - Centro Oncológico Gallego José Antonio Quiroga y Piñeiro, Servicio de Oncologia, A Coruña
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital de San Pedro de Alcantara, Cáceres
  - Hospital Universitari Arnau de Vilanova de Lleida; Servicio de Oncologia, Lleida
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen de Arrixaca; Servicio de Oncologia, Murcia
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Turkey (Türkiye) (4):
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Ankara
  - Ankara City Hospital, Ankara
  - Ege Uni Medical Faculty Hospital; Oncology Dept, Izmir
  - Inonu University Medical Faculty Turgut Ozal Medical Center Medical Oncology Department, Malatya
- United Kingdom (7):
  - Brighton and Sussex Univ Hosp, Brighton
  - University Hospital coventry; Oncology Department, Coventry
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Queen Elizabeth Hospital, London
  - Queen Alexandra Hospital, Portsmouth, Portsmouth
  - Scarborough General Hospital, Scarborough
  - Weston Park Hospital; Cancer Clinical Trials Centre, Sheffield

REFERENCES:
- [Derived] Rimawi M, Ferrero JM, de la Haba-Rodriguez J, Poole C, De Placido S, Osborne CK, Hegg R, Easton V, Wohlfarth C, Arpino G; PERTAIN Study Group. First-Line Trastuzumab Plus an Aromatase Inhibitor, With or Without Pertuzumab, in Human Epidermal Growth Factor Receptor 2-Positive and Hormone Receptor-Positive Metastatic or Locally Advanced Breast Cancer (PERTAIN): A Randomized, Open-Label Phase II Trial. J Clin Oncol. 2018 Oct 1;36(28):2826-2835. doi: 10.1200/JCO.2017.76.7863. Epub 2018 Aug 14. PMID 30106636

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 258 participants were enrolled in the study.
Groups:
- Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy: Participants received pertuzumab at a loading dose of 840 mg followed by 420 mg along with trastuzumab at a loading dose of 8 mg/kg of body weight followed by 6 mg/kg of body weight on Day 1 or Day 2 of each 3-weekly cycle until disease progression, unacceptable toxicity, withdrawal of consent, or death, or the predefined end of study whichever occurred first. Participants also received an aromatase inhibitor (AI), orally as per product labeling (anastrozole: 1 mg once daily or letrozole: 2.5 mg once daily). Participants receiving induction chemotherapy up to the first 18-24 weeks of the treatment period were to receive a taxane (docetaxel every 3 weeks or paclitaxel weekly), administered in line with the respective product labeling.
- Arm B: Trastuzumab + AI +/- Chemotherapy: Participants received trastuzumab at a loading dose of 8 mg/kg of body weight followed by 6 mg/kg of body weight on Day 1 or Day 2 of each 3-weekly cycle until disease progression, unacceptable toxicity, withdrawal of consent, or death, or the predefined end of study whichever occurred first. Participants also received an aromatase inhibitor (AI), orally as per product labeling (anastrozole: 1 mg once daily or letrozole: 2.5 mg once daily). Participants receiving induction chemotherapy up to the first 18-24 weeks of the treatment period were to receive a taxane (docetaxel every 3 weeks or paclitaxel weekly), administered in line with the respective product labeling.
Period: Overall Study
Arm/Group | Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy | Arm B: Trastuzumab + AI +/- Chemotherapy
Started (Intent-to-Treat (ITT) Population) | 129 | 129
Received at Least One Dose of Study Drug (Safety Population) | 127 | 124
Entered Follow-Up (Post-Treatment) | 120 | 116
Completed | 0 | 0
Not Completed | 129 | 129
Not completed — Withdrawal by Subject | 20 | 17
Not completed — Lost to Follow-up | 2 | 10
Not completed — Death | 63 | 57
Not completed — Study Termination by Sponsor | 36 | 36
Not completed — Reason Not Specified | 8 | 9

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy | Arm B: Trastuzumab + AI +/- Chemotherapy | Total
Number analyzed (Participants) | 129 | 129 | 258
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (10.85) | 62.3 (11.54) | 61.6 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 129 | 258
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 10 | 18 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 104 | 93 | 197
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 12 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 45 | 40 | 85
  Chinese | 0 | 0 | 0
  Indian (Indian subcontinent) | 10 | 16 | 26
  Japanese | 0 | 1 | 1
  Mixed Ethnicity | 0 | 0 | 0
  Other | 63 | 60 | 123
  Missing | 11 | 12 | 23
Number of Participants by Induction Chemotherapy and Prior Adjuvant Hormone Therapy [Count of Participants; unit: Participants] — Participants were stratified at randomization according to the following factors: -Chosen to receive induction chemotherapy? (Yes vs. No); -Time since adjuvant hormone therapy (<12 months vs. ≥12 months), or no prior hormone therapy. Population: All 258 participants who were enrolled on this study are accounted for between the induction chemotherapy categories (yes vs. no).
  Participants
    Induction Chemotherapy - Yes: number analyzed (Participants) | 75 | 73 | 148
    Induction Chemotherapy - Yes: <12 Months Since Hormone Therapy | 12 | 12 | 24
    Induction Chemotherapy - Yes: ≥12 Months Since Hormone Therapy | 24 | 23 | 47
    Induction Chemotherapy - Yes: No Prior Hormone Therapy | 39 | 38 | 77
    Induction Chemotherapy - No: number analyzed (Participants) | 54 | 56 | 110
    Induction Chemotherapy - No: <12 Months Since Hormone Therapy | 12 | 12 | 24
    Induction Chemotherapy - No: ≥12 Months Since Hormone Therapy | 18 | 19 | 37
    Induction Chemotherapy - No: No Prior Hormone Therapy | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time from randomization until the first radiographically documented progression of disease or death from any cause, whichever occurred first (either during study treatment or during follow-up). Progression of disease was evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1 and is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum of target lesion diameters must also demonstrate an absolute increase of at least 5 mm (Note: the appearance of one or more new lesions is also considered progression). Participants with no PFS events were censored at the time of the last evaluable tumor assessment. The primary analysis of PFS was planned to be performed when a total of 165 PFS events had occurred, and the final analysis after at least 60 months follow-up.
Time Frame: Median [full range] of follow-up time on study for: Primary Analysis: 31.7 [0.0-44.3] months vs. 30.4 [0.0-45.8] months in Arm A vs. Arm B; Final Analysis: 73.20 [0.03-88.34] months vs. 71.06 [0.03-88.97] months in Arm A vs. Arm B
Population: Intent-to-Treat (ITT) population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy | Arm B: Trastuzumab + AI +/- Chemotherapy
Number analyzed (Participants) | 129 | 129
months
  Primary Analysis | 18.89 [14.09 to 27.66] | 15.80 [11.04 to 18.56]
  Final Analysis | 20.63 [14.39 to 28.35] | 15.80 [11.04 to 18.66]
Statistical Analysis 1: Comparison: Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy vs Arm B: Trastuzumab + AI +/- Chemotherapy; Primary Analysis. Log Rank tested the following: Null Hypothesis (H0): the distribution of the PFS time was the same in Arms A & B; The Alternative Hypothesis (H1): the distribution of the PFS time was different in Arms A & B. A Cox proportional hazards model tested the HR. If the HR of investigational arm (Arm A) compared with control arm (Arm B) with respect to PFS was assumed to be constant over time (λ) then the null (H0) and alternative hypotheses (H1) were: H0: λ =1; H1: λ ≠1; Test type: Superiority; p = 0.0070, Log Rank — Test was performed at 2-sided alpha of 5%; Stratified log-rank test based upon Kaplan-Meier including induction chemotherapy and prior adjuvant hormone therapy stratification factors; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.48 to 0.89] — Hazard ratio comparing Arm A vs. B from stratified Cox proportional hazards model including stratification factors
Statistical Analysis 2: Comparison: Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy vs Arm B: Trastuzumab + AI +/- Chemotherapy; Final Analysis; Test type: Other — Exploratory; p = 0.0059, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.50 to 0.89] — Hazard ratio comparing Arm A vs. B from stratified Cox proportional hazards model including stratification factors

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from the date of randomization to the date of death, regardless of the cause of death. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last study medication (pertuzumab, trastuzumab, AI or induction chemotherapy), and participants with no post-baseline information were censored at the date of randomization. The primary analysis of OS was planned to be performed at the same time as for PFS (when a total of 165 PFS events had occurred), and the final analysis was planned after at least 60 months follow-up for all participants.
Time Frame: as for outcome 1
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy | Arm B: Trastuzumab + AI +/- Chemotherapy
Number analyzed (Participants) | 129 | 129
Months
  Primary Analysis | NA [NA to NA] — Median and lower and upper limits of the 95% confidence interval were not reached because not enough events had occurred at the time of analysis. | NA [41.40 to NA] — Median and upper limit of the 95% confidence interval were not reached because not enough events had occurred at the time of analysis.
  Final Analysis | 60.16 [47.21 to 79.01] | 57.17 [45.44 to NA] — Upper limit of 95% confidence interval was not reached because not enough events had occurred the time of analysis.
Statistical Analysis 1: Comparison: Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy vs Arm B: Trastuzumab + AI +/- Chemotherapy; Primary Analysis. This study was not powered for overall survival (OS), so adequately powered statistical testing for this outcome measure was not possible; Test type: Other — Exploratory; p = 0.5850, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.69 to 1.91] — Hazard ratio comparing Arm A vs. B from stratified Cox proportional hazards model including stratification factors
Statistical Analysis 2: Comparison: Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy vs Arm B: Trastuzumab + AI +/- Chemotherapy; Final Analysis. This study was not powered for overall survival (OS), so adequately powered statistical testing for this outcome measure was not possible; Test type: Other — Exploratory; p = 0.7833, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.73 to 1.52] — Hazard ratio comparing Arm A vs. B from stratified Cox proportional hazards model including stratification factors

3. Secondary Outcome: Overall Response Rate (ORR)
Description: The overall response rate (ORR) was defined as the percentage of participants with best (confirmed) overall response (BOR) of either complete response (CR) or partial response (PR) from start of study treatment until progressive disease (PD)/recurrence or death, as assessed by the investigator according to RECIST version 1.1. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm; PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference baseline sum diameters; stable disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Participants needed to have two consecutive assessments of PR or CR at least 4 weeks apart to be a responder. Analysis of this outcome measure was only planned to occur at the time of primary analysis.
Time Frame: Median [full range] of follow-up time on study for Primary Analysis: 31.7 [0.0-44.3] months vs. 30.4 [0.0-45.8] months in Arm A vs. Arm B
Population: ITT population included all randomized participants. Only participants with measurable disease at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy | Arm B: Trastuzumab + AI +/- Chemotherapy
Number analyzed (Participants) | 109 | 106
percentage of participants
  ORR (CR + PR) | 63.3 [53.5 to 72.3] | 55.7 [45.7 to 65.3]
  Non-responders (SD + PD + NE) | 36.7 [27.7 to 46.5] | 44.3 [34.7 to 54.3]
  Complete Response (CR) | 7.3 [3.2 to 14.0] | 0.9 [0.0 to 5.1]
  Partial Response (PR) | 56.0 [46.1 to 65.5] | 54.7 [44.8 to 64.4]
  Stable Disease (SD) | 26.6 [18.6 to 35.9] | 27.4 [19.1 to 36.9]
  Progressive Disease (PD) | 5.5 [2.0 to 11.6] | 12.3 [6.7 to 20.1]
  Not Evaluable (NE) | 4.5 [1.5 to 10.4] | 4.7 [1.5 to 10.7]
Statistical Analysis 1: Comparison: Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy vs Arm B: Trastuzumab + AI +/- Chemotherapy; ORR for Arm A vs Arm B; Test type: Superiority; p = 0.2537, Chi-squared — Test was performed at 2-sided alpha of 5%. There was no multiplicity adjustment; Difference in ORR = 7.6, 95% CI 2-sided [-6.0 to 21.3]

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical Benefit Rate (CBR) was defined as the percentage of participants with best (confirmed) partial response (PR) or complete response (CR) or stable disease (SD) for at least 6 months. According to RECIST version 1.1, CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm; PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Analysis of this outcome measure was only planned to occur at the time of primary analysis.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy | Arm B: Trastuzumab + AI +/- Chemotherapy
Number analyzed (Participants) | 109 | 106
percentage of participants
  CBR (CR + PR + SD for ≥6 Months) | 68.8 [59.2 to 77.3] | 67.0 [57.2 to 75.8]
  Complete Response (CR) | 7.3 [3.2 to 14.0] | 0.9 [0.0 to 5.1]
  Partial Response (PR) | 56.0 [46.1 to 65.5] | 54.7 [44.8 to 64.4]
  Stable Disease (SD) for ≥6 Months | 5.5 [2.0 to 11.6] | 11.3 [6.0 to 18.9]
Statistical Analysis 1: Comparison: Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy vs Arm B: Trastuzumab + AI +/- Chemotherapy; CBR for Arm A vs. Arm B; Test type: Superiority; p = 0.7743, Chi-squared — Test was performed at 2-sided alpha of 5%. There was no multiplicity adjustment; Difference in CBR = 1.8, 95% CI 2-sided [-11.2 to 14.8]

5. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) was defined as the period from the date of initial confirmed partial response (PR) or complete response (CR) until the date of progressive disease or death from any cause. According to RECIST version 1.1, CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm; PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Participants with no documented progression after CR or PR were censored at the last date at which they were known to have had the CR or PR, respectively. The primary analysis of DOR was planned to be performed at the same time as for PFS (when a total of 165 PFS events had occurred), and the final analysis was planned after at least 60 months follow-up for all participants.
Time Frame: as for outcome 1
Population: ITT population included all randomized participants. Only participants who had measurable disease at baseline and were responders (CR or PR) were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy | Arm B: Trastuzumab + AI +/- Chemotherapy
Number analyzed (Participants) | 69 | 61
months
  Primary Analysis: number analyzed (Participants) | 69 | 59
  Primary Analysis | 27.10 [14.13 to NA] — Upper limit of the 95% confidence interval was not reached because not enough events had occurred at the time of analysis. | 15.11 [12.09 to 20.96]
  Final Analysis | 27.40 [15.24 to 44.35] | 16.36 [12.09 to 20.96]
Statistical Analysis 1: Comparison: Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy vs Arm B: Trastuzumab + AI +/- Chemotherapy; Primary Analysis. Log Rank tested the following: Null Hypothesis (H0): the distribution of the DOR time was the same in Arms A & B; The Alternative Hypothesis (H1): the distribution of the DOR time was different in Arms A & B. A Cox proportional hazards model tested the HR. If the HR of investigational arm (Arm A) compared with control arm (Arm B) with respect to DOR was assumed to be constant over time (λ) then the null (H0) and alternative hypotheses (H1) were: H0: λ =1; H1: λ ≠1; Test type: Superiority; p = 0.0181, Log Rank — Test was performed at 2-sided alpha of 5%; Log-rank test from unstratified analysis based upon Kaplan-Meier approach. There was no multiplicity adjustment; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.36 to 0.91] — Hazard ratio from stratified Cox proportional hazards model including stratification factors of induction chemotherapy and prior adjuvant hormone therapy
Statistical Analysis 2: Comparison: Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy vs Arm B: Trastuzumab + AI +/- Chemotherapy; Final Analysis; Test type: Other — Exploratory; p = 0.0205, Log Rank; Log-rank test from unstratified analysis based upon Kaplan-Meier approach. There was no multiplicity adjustment; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.41 to 0.93] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Time to Response (TTR)
Description: Time to Response (TTR) was defined as the time from the date of randomization to the date of first complete response (CR) or partial response (PR). According to RECIST version 1.1, CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm; PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. For participants who did not have a confirmed response, a censored TTR was calculated at the date of the last adequate tumor assessment. If no tumor assessment is performed for the participant (or all post-baseline assessments are not evaluable or PD) the censoring day would be set to day 1 (date of randomization). Analysis of this outcome measure was only planned to occur at the time of primary analysis.
Time Frame: as for outcome 3
Population: ITT population included all randomized participants. Only participants with measurable disease at baseline were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy | Arm B: Trastuzumab + AI +/- Chemotherapy
Number analyzed (Participants) | 109 | 106
months | 2.53 [2.10 to 4.37] | 3.91 [2.10 to 4.17]
Statistical Analysis 1: Comparison: Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy vs Arm B: Trastuzumab + AI +/- Chemotherapy; Log Rank tested the following: Null Hypothesis (H0): the distribution of the TTR time was the same in Arms A & B; The Alternative Hypothesis (H1): the distribution of the TTR time was different in Arms A & B. A Cox proportional hazards model tested the HR. If the HR of investigational arm (Arm A) compared with control arm (Arm B) with respect to TTR was assumed to be constant over time (λ) then the null (H0) and alternative hypotheses (H1) were: H0: λ =1; H1: λ ≠1; Test type: Superiority; p = 0.5597, Log Rank — Test was performed at 2-sided alpha of 5%; The log-rank test from unstratified analysis was based upon Kaplan-Meier approach. There was no multiplicity adjustment; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.78 to 1.57] — Hazard ratio from stratified Cox proportional hazards model including the induction chemotherapy and prior adjuvant hormone therapy stratification factors

7. Secondary Outcome: Change From Baseline in Health-Related Quality of Life as Determined by European Quality of Life 5-Dimension (EQ-5D) Visual Analog Scale (VAS) Scores
Description: The EQ-5D VAS is a participant-rated questionnaire to assess health-related quality of life (QoL) in terms of a single index value. The VAS component rates current health state on a scale from 0 mm (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline and every 3 cycles until treatment discontinuation (up to Cycle 120; 1 cycle is 21 days)
Population: ITT population included all randomized participants. The number analyzed only included those who had a non-missing assessment for a specified time point.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy | Arm B: Trastuzumab + AI +/- Chemotherapy
Number analyzed (Participants) | 129 | 129
unit on a scale
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 98 | 101
  Baseline (BL) - Value at Visit | 73.0 (19.34) | 72.8 (18.83)
  Change from BL at Cycle 3: number analyzed (Participants) | 87 | 87
  Change from BL at Cycle 3 | 3.3 (14.90) | 1.9 (15.67)
  Change from BL at Cycle 6: number analyzed (Participants) | 82 | 75
  Change from BL at Cycle 6 | 3.5 (18.91) | 0.5 (13.63)
  Change from BL at Cycle 9: number analyzed (Participants) | 68 | 66
  Change from BL at Cycle 9 | 5.3 (18.80) | 2.1 (15.20)
  Change from BL at Cycle 12: number analyzed (Participants) | 58 | 52
  Change from BL at Cycle 12 | 10.7 (17.91) | 4.0 (15.34)
  Change from BL at Cycle 15: number analyzed (Participants) | 54 | 50
  Change from BL at Cycle 15 | 9.1 (17.25) | 1.4 (22.16)
  Change from BL at Cycle 18: number analyzed (Participants) | 47 | 43
  Change from BL at Cycle 18 | 7.5 (12.85) | 3.5 (15.76)
  Change from BL at Cycle 21: number analyzed (Participants) | 44 | 39
  Change from BL at Cycle 21 | 5.8 (13.68) | 3.5 (19.70)
  Change from BL at Cycle 24: number analyzed (Participants) | 39 | 38
  Change from BL at Cycle 24 | 6.2 (14.30) | 3.2 (16.66)
  Change from BL at Cycle 27: number analyzed (Participants) | 35 | 34
  Change from BL at Cycle 27 | 7.5 (14.01) | 3.9 (22.00)
  Change from BL at Cycle 30: number analyzed (Participants) | 33 | 29
  Change from BL at Cycle 30 | 8.3 (14.25) | 4.9 (16.98)
  Change from BL at Cycle 33: number analyzed (Participants) | 34 | 24
  Change from BL at Cycle 33 | 5.1 (14.70) | 4.3 (15.59)
  Change from BL at Cycle 36: number analyzed (Participants) | 30 | 21
  Change from BL at Cycle 36 | 7.3 (15.19) | 5.9 (15.13)
  Change from BL at Cycle 39: number analyzed (Participants) | 30 | 18
  Change from BL at Cycle 39 | 8.1 (16.33) | 2.4 (29.68)
  Change from BL at Cycle 42: number analyzed (Participants) | 25 | 15
  Change from BL at Cycle 42 | 6.4 (19.18) | 9.0 (17.55)
  Change from BL at Cycle 45: number analyzed (Participants) | 22 | 14
  Change from BL at Cycle 45 | 9.7 (15.01) | 9.9 (19.52)
  Change from BL at Cycle 48: number analyzed (Participants) | 19 | 13
  Change from BL at Cycle 48 | 8.8 (12.50) | 6.8 (17.22)
  Change from BL at Cycle 51: number analyzed (Participants) | 18 | 13
  Change from BL at Cycle 51 | 7.2 (14.81) | 9.1 (19.11)
  Change from BL at Cycle 54: number analyzed (Participants) | 16 | 12
  Change from BL at Cycle 54 | 4.7 (23.48) | 7.6 (17.85)
  Change from BL at Cycle 57: number analyzed (Participants) | 16 | 11
  Change from BL at Cycle 57 | 6.8 (18.08) | 10.5 (16.81)
  Change from BL at Cycle 60: number analyzed (Participants) | 16 | 11
  Change from BL at Cycle 60 | 8.2 (15.88) | 10.9 (18.27)
  Change from BL at Cycle 63: number analyzed (Participants) | 16 | 10
  Change from BL at Cycle 63 | 4.0 (20.88) | 8.8 (14.64)
  Change from BL at Cycle 66: number analyzed (Participants) | 14 | 8
  Change from BL at Cycle 66 | 10.4 (16.92) | 4.1 (15.69)
  Change from BL at Cycle 69: number analyzed (Participants) | 13 | 7
  Change from BL at Cycle 69 | 7.5 (17.35) | 5.0 (16.77)
  Change from BL at Cycle 72: number analyzed (Participants) | 13 | 8
  Change from BL at Cycle 72 | 6.2 (16.10) | 5.8 (16.10)
  Change from BL at Cycle 75: number analyzed (Participants) | 11 | 7
  Change from BL at Cycle 75 | 8.6 (19.12) | 5.1 (15.50)
  Change from BL at Cycle 78: number analyzed (Participants) | 11 | 7
  Change from BL at Cycle 78 | 12.8 (17.45) | 6.9 (14.58)
  Change from BL at Cycle 81: number analyzed (Participants) | 11 | 6
  Change from BL at Cycle 81 | 11.5 (18.39) | 8.0 (14.76)
  Change from BL at Cycle 84: number analyzed (Participants) | 11 | 6
  Change from BL at Cycle 84 | 11.2 (19.71) | 1.3 (18.13)
  Change from BL at Cycle 87: number analyzed (Participants) | 11 | 4
  Change from BL at Cycle 87 | 11.2 (18.17) | -3.0 (11.22)
  Change from BL at Cycle 90: number analyzed (Participants) | 11 | 4
  Change from BL at Cycle 90 | 10.9 (18.28) | -3.0 (12.36)
  Change from BL at Cycle 93: number analyzed (Participants) | 11 | 5
  Change from BL at Cycle 93 | 7.1 (15.43) | 6.6 (13.89)
  Change from BL at Cycle 96: number analyzed (Participants) | 8 | 5
  Change from BL at Cycle 96 | 7.5 (16.04) | 8.6 (12.64)
  Change from BL at Cycle 99: number analyzed (Participants) | 9 | 5
  Change from BL at Cycle 99 | 4.4 (17.22) | 5.6 (16.71)
  Change from BL at Cycle 102: number analyzed (Participants) | 8 | 3
  Change from BL at Cycle 102 | 5.6 (16.35) | 10.0 (17.32)
  Change from BL at Cycle 105: number analyzed (Participants) | 8 | 1
  Change from BL at Cycle 105 | 4.4 (16.35) | 0.0 (NA) — Standard deviation could not be calculated using data from a single participant.
  Change from BL at Cycle 108: number analyzed (Participants) | 7 | 1
  Change from BL at Cycle 108 | 4.0 (14.39) | 0.0 (NA) — Standard deviation could not be calculated using data from a single participant.
  Change from BL at Cycle 111: number analyzed (Participants) | 4 | 0
  Change from BL at Cycle 111 | 3.3 (21.50) |
  Change from BL at Cycle 114: number analyzed (Participants) | 4 | 0
  Change from BL at Cycle 114 | -1.3 (17.97) |
  Change from BL at Cycle 117: number analyzed (Participants) | 1 | 0
  Change from BL at Cycle 117 | -5.0 (NA) — Standard deviation could not be calculated using data from a single participant. |
  Change from BL at Cycle 120: number analyzed (Participants) | 1 | 0
  Change from BL at Cycle 120 | -5.0 (NA) — Standard deviation could not be calculated using data from a single participant. |

8. Secondary Outcome: Overview of the Number of Participants With Adverse Events, Severity Determined According to NCI-CTCAE Version 4.03
Description: All adverse events (AEs) occurring during the study and until the post-treatment safety follow-up visit approximately 28 days after last study medication were recorded; thereafter, only study drug-related serious adverse events (SAEs) continued to be collected. The investigator graded all AEs for severity per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.03; if not listed, the AE was assessed as follows: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening/disabling; Grade 5 = death. The investigator determined whether an AE was related to study drug and independently assessed severity and seriousness of each AE. AEs suggestive of congestive heart failure (CHF) were identified by the SMQ (wide) "Cardiac Failure" with a status of "serious", which included the preferred terms cardiac failure, left ventricular dysfunction, and pulmonary oedema.
Time Frame: From Baseline until the end of post-treatment follow-up (up to 89 months)
Population: Safety population: included all participants who had received at least 1 dose of any study medication assigned to treatment arms as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy | Arm B: Trastuzumab + AI +/- Chemotherapy
Number analyzed (Participants) | 127 | 124
Participants
  Any Adverse Event (AE) | 122 | 122
  Any AE, Grade ≥3 | 72 | 51
  Any Serious Adverse Event (SAE), Grade ≥3 | 35 | 22
  Any AE, Grade 5 | 1 | 1
  Any SAE | 46 | 28
  SAE Related to Pertuzumab | 10 | NA — None of the participants in Arm B were treated with pertuzumab.
  SAE Related to Trastuzumab | 9 | 2
  SAE Related to Docetaxel: number analyzed (Participants) | 74 | 69
  SAE Related to Docetaxel | 6 | 4
  SAE Related to Paclitaxel: number analyzed (Participants) | 74 | 69
  SAE Related to Paclitaxel | 3 | 0
  Any AE Leading to Discontinuation of Any Treatment | 20 | 10
  Any AE Leading to Pertuzumab Discontinuation | 16 | NA — None of the participants in Arm B were treated with pertuzumab.
  Any AE Leading to Trastuzumab Discontinuation | 16 | 6
  Any AE Leading to Interruption of Any Treatment | 59 | 26
  Any AE Leading to Pertuzumab Interruption | 44 | NA — None of the participants in Arm B were treated with pertuzumab.
  Any AE Leading to Trastuzumab Interruption | 48 | 16
  Any AE Related to Pertuzumab | 82 | NA — None of the participants in Arm B were treated with pertuzumab.
  Any AE Related to Trastuzumab | 81 | 62
  AE Suggestive of Congestive Heart Failure | 5 | 1

9. Secondary Outcome: Number of Participants Who Died Over the Course of the Study by Reported Cause of Death and Time of Death Relative to First or Last Dose of Study Treatment
Description: The causes of death over the course of the study, regardless of whether the death was related to study treatment, are listed by preferred term according to the Medical Dictionary for Regulatory Activities (MedDRA), version 22.1.
Time Frame: From Baseline until the end of post-treatment follow-up (up to 89 months)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy | Arm B: Trastuzumab + AI +/- Chemotherapy
Number analyzed (Participants) | 127 | 124
Participants
  Total Number of Deaths | 62 | 57
  Deaths Related to Any Study Treatment | 0 | 0
  Cause of Death: Cardiac Arrest | 1 | 0
  Cause of Death: Craniocerebral Injury | 1 | 0
  Cause of Death: Dyspnoea | 1 | 0
  Cause of Death: High-grade B-cell Lymphoma | 1 | 0
  Cause of Death: Sudden Death | 0 | 1
  Cause of Death: Unevaluable Event | 2 | 1
  Cause of Death: Progressive Disease | 56 | 55
  Total Deaths Within 30 Days After First Dose | 0 | 0
  Total Deaths Within 28 Days After Last Dose | 1 | 2
  Total Deaths Within 60 Days After Last Dose | 2 | 4

10. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) Values Over the Course of the Study
Description: Left ventricular ejection fraction (LVEF) is the measurement of how much blood is being pumped out of the left ventricle of the heart (the main pumping chamber) with each contraction. A normal LVEF ranges from 55% to 70%, as measured by echocardiogram or multiple-gated acquisition (MUGA) scan. All participants must have had a baseline LVEF of at least (≥)50% to enroll in the study; patients with clinically significant cardiovascular disease or baseline LVEF below 50% were not eligible for this study.
Time Frame: Baseline and every 3 cycles until treatment discontinuation (up to Cycle 120; 1 cycle is 21 days)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage points of LVEF
Arm/Group | Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy | Arm B: Trastuzumab + AI +/- Chemotherapy
Number analyzed (Participants) | 127 | 124
Percentage points of LVEF
  Baseline (BL) - Absolute LVEF at Visit: number analyzed (Participants) | 127 | 123
  Baseline (BL) - Absolute LVEF at Visit | 63.8 (6.23) | 63.9 (6.12)
  Change from BL at Cycle 3: number analyzed (Participants) | 114 | 114
  Change from BL at Cycle 3 | -1.0 (6.25) | -1.4 (6.23)
  Change from BL at Cycle 6: number analyzed (Participants) | 101 | 101
  Change from BL at Cycle 6 | -2.3 (6.66) | -1.3 (6.03)
  Change from BL at Cycle 9: number analyzed (Participants) | 87 | 84
  Change from BL at Cycle 9 | -2.5 (6.80) | -2.2 (6.52)
  Change from BL at Cycle 12: number analyzed (Participants) | 75 | 69
  Change from BL at Cycle 12 | -2.4 (8.05) | -2.8 (6.99)
  Change from BL at Cycle 15: number analyzed (Participants) | 64 | 61
  Change from BL at Cycle 15 | -2.9 (8.67) | -2.5 (6.94)
  Change from BL at Cycle 18: number analyzed (Participants) | 62 | 54
  Change from BL at Cycle 18 | -1.9 (6.42) | -1.3 (6.19)
  Change from BL at Cycle 21: number analyzed (Participants) | 53 | 48
  Change from BL at Cycle 21 | -1.1 (6.01) | -1.1 (6.64)
  Change from BL at Cycle 24: number analyzed (Participants) | 52 | 46
  Change from BL at Cycle 24 | -2.1 (6.82) | -0.6 (6.19)
  Change from BL at Cycle 27: number analyzed (Participants) | 46 | 39
  Change from BL at Cycle 27 | -1.6 (5.05) | -1.3 (5.87)
  Change from BL at Cycle 30: number analyzed (Participants) | 43 | 34
  Change from BL at Cycle 30 | -1.4 (5.20) | -0.3 (6.03)
  Change from BL at Cycle 33: number analyzed (Participants) | 44 | 28
  Change from BL at Cycle 33 | -2.8 (5.60) | 1.2 (6.71)
  Change from BL at Cycle 36: number analyzed (Participants) | 37 | 24
  Change from BL at Cycle 36 | -2.5 (5.50) | -0.2 (5.41)
  Change from BL at Cycle 39: number analyzed (Participants) | 38 | 23
  Change from BL at Cycle 39 | -2.6 (5.72) | 1.4 (4.87)
  Change from BL at Cycle 42: number analyzed (Participants) | 35 | 18
  Change from BL at Cycle 42 | -2.1 (5.91) | 1.9 (6.12)
  Change from BL at Cycle 45: number analyzed (Participants) | 31 | 17
  Change from BL at Cycle 45 | -1.0 (5.54) | 3.0 (5.27)
  Change from BL at Cycle 48: number analyzed (Participants) | 28 | 18
  Change from BL at Cycle 48 | -3.3 (6.56) | -0.2 (7.50)
  Change from BL at Cycle 51: number analyzed (Participants) | 27 | 18
  Change from BL at Cycle 51 | -1.4 (5.82) | 1.0 (4.19)
  Change from BL at Cycle 54: number analyzed (Participants) | 26 | 13
  Change from BL at Cycle 54 | -1.3 (6.17) | -1.0 (6.23)
  Change from BL at Cycle 57: number analyzed (Participants) | 26 | 15
  Change from BL at Cycle 57 | -1.7 (6.43) | 0.8 (5.68)
  Change from BL at Cycle 60: number analyzed (Participants) | 25 | 14
  Change from BL at Cycle 60 | -2.5 (5.54) | -0.9 (3.91)
  Change from BL at Cycle 63: number analyzed (Participants) | 26 | 14
  Change from BL at Cycle 63 | -2.1 (6.10) | 0.8 (5.99)
  Change from BL at Cycle 66: number analyzed (Participants) | 22 | 13
  Change from BL at Cycle 66 | -2.9 (7.80) | -0.4 (5.17)
  Change from BL at Cycle 69: number analyzed (Participants) | 19 | 9
  Change from BL at Cycle 69 | -2.1 (7.23) | -1.5 (7.68)
  Change from BL at Cycle 72: number analyzed (Participants) | 18 | 12
  Change from BL at Cycle 72 | -3.0 (4.97) | -1.0 (5.75)
  Change from BL at Cycle 75: number analyzed (Participants) | 17 | 12
  Change from BL at Cycle 75 | -3.3 (6.59) | -1.1 (6.97)
  Change from BL at Cycle 78: number analyzed (Participants) | 17 | 9
  Change from BL at Cycle 78 | -3.3 (5.58) | -1.1 (7.82)
  Change from BL at Cycle 81: number analyzed (Participants) | 17 | 9
  Change from BL at Cycle 81 | -2.9 (6.83) | -2.6 (6.00)
  Change from BL at Cycle 84: number analyzed (Participants) | 15 | 9
  Change from BL at Cycle 84 | -2.5 (7.66) | -4.5 (3.59)
  Change from BL at Cycle 87: number analyzed (Participants) | 15 | 8
  Change from BL at Cycle 87 | -3.8 (5.76) | -1.4 (5.12)
  Change from BL at Cycle 90: number analyzed (Participants) | 16 | 7
  Change from BL at Cycle 90 | -2.4 (7.69) | 0.4 (6.77)
  Change from BL at Cycle 93: number analyzed (Participants) | 14 | 7
  Change from BL at Cycle 93 | -1.8 (6.57) | -3.9 (6.00)
  Change from BL at Cycle 96: number analyzed (Participants) | 12 | 7
  Change from BL at Cycle 96 | -0.7 (7.45) | -3.2 (5.50)
  Change from BL at Cycle 99: number analyzed (Participants) | 11 | 7
  Change from BL at Cycle 99 | -3.4 (5.78) | -2.8 (8.41)
  Change from BL at Cycle 102: number analyzed (Participants) | 13 | 5
  Change from BL at Cycle 102 | -1.3 (6.12) | -1.6 (9.68)
  Change from BL at Cycle 105: number analyzed (Participants) | 12 | 3
  Change from BL at Cycle 105 | -0.4 (7.05) | -2.0 (12.17)
  Change from BL at Cycle 108: number analyzed (Participants) | 9 | 3
  Change from BL at Cycle 108 | -3.4 (5.32) | -3.3 (8.33)
  Change from BL at Cycle 111: number analyzed (Participants) | 4 | 1
  Change from BL at Cycle 111 | -6.3 (5.91) | -5.5 (NA) — Standard deviation could not be calculated with data from a single participant.
  Change from BL at Cycle 114: number analyzed (Participants) | 4 | 1
  Change from BL at Cycle 114 | -4.0 (5.35) | -1.4 (NA) — Standard deviation could not be calculated with data from a single participant.
  Change from BL at Cycle 117: number analyzed (Participants) | 1 | 0
  Change from BL at Cycle 117 | -11.0 (NA) — Standard deviation could not be calculated with data from a single participant. |
  Change from BL at Cycle 120: number analyzed (Participants) | 1 | 0
  Change from BL at Cycle 120 | -11.0 (NA) — Standard deviation could not be calculated with data from a single participant. |

ADVERSE EVENTS:
Time Frame: From Baseline until end of post-treatment follow-up (up to 89 months)
Description: All adverse events that occurred during the study and until the post-treatment safety follow-up visit approximately 28 days after last study medication were to be recorded. Thereafter, only serious adverse events thought to be related to study drug were collected.
Arm/Group | Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy | Arm B: Trastuzumab + AI +/- Chemotherapy
All-Cause Mortality (participants affected / at risk) | 63/129 | 57/129
Serious Adverse Events (participants affected / at risk) | 46/127 | 28/124
Other Adverse Events (participants affected / at risk) | 120/127 | 116/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy (N=127) | Arm B: Trastuzumab + AI +/- Chemotherapy (N=124)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 4 (4) | 0 (0)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal haemorrhage (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 3 (3) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 2 (2)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 6 (7) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenoid cystic carcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
High-grade B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Colostomy closure (Surgical and medical procedures) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour exudation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Pertuzumab + Trastuzumab + AI +/- Chemotherapy (N=127) | Arm B: Trastuzumab + AI +/- Chemotherapy (N=124)
Anaemia (Blood and lymphatic system disorders) | 28 (53) | 18 (30)
Neutropenia (Blood and lymphatic system disorders) | 11 (14) | 13 (23)
Lacrimation increased (Eye disorders) | 9 (9) | 7 (8)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 16 (18)
Abdominal pain upper (Gastrointestinal disorders) | 12 (17) | 6 (6)
Constipation (Gastrointestinal disorders) | 18 (27) | 19 (25)
Diarrhoea (Gastrointestinal disorders) | 70 (213) | 45 (88)
Dyspepsia (Gastrointestinal disorders) | 8 (9) | 9 (11)
Nausea (Gastrointestinal disorders) | 47 (68) | 34 (56)
Stomatitis (Gastrointestinal disorders) | 17 (24) | 11 (22)
Vomiting (Gastrointestinal disorders) | 31 (42) | 21 (33)
Asthenia (General disorders) | 39 (76) | 32 (77)
Chest Pain (General disorders) | 9 (11) | 9 (11)
Chills (General disorders) | 8 (8) | 7 (8)
Fatigue (General disorders) | 21 (33) | 25 (43)
Influenza like illness (General disorders) | 10 (17) | 7 (10)
Mucosal inflammation (General disorders) | 14 (20) | 13 (15)
Oedema peripheral (General disorders) | 34 (53) | 23 (34)
Pyrexia (General disorders) | 17 (22) | 13 (14)
Influenza (Infections and infestations) | 6 (10) | 7 (12)
Nasopharyngitis (Infections and infestations) | 13 (21) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 13 (36) | 15 (23)
Urinary tract infection (Infections and infestations) | 17 (25) | 16 (20)
Ejection fraction decreased (Investigations) | 13 (19) | 8 (9)
Weight decreased (Investigations) | 14 (16) | 11 (12)
Weight increased (Investigations) | 11 (13) | 5 (10)
Decreased appetite (Metabolism and nutrition disorders) | 23 (27) | 10 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 (60) | 31 (49)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (29) | 21 (27)
Bone pain (Musculoskeletal and connective tissue disorders) | 16 (25) | 10 (12)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 (17) | 5 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 11 (13) | 4 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 6 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (16) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 (44) | 16 (23)
Dizziness (Nervous system disorders) | 21 (32) | 12 (12)
Headache (Nervous system disorders) | 22 (33) | 14 (24)
Neuropathy peripheral (Nervous system disorders) | 18 (26) | 17 (19)
Paraesthesia (Nervous system disorders) | 13 (19) | 11 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (12) | 9 (9)
Anxiety (Psychiatric disorders) | 14 (15) | 5 (6)
Depression (Psychiatric disorders) | 13 (14) | 5 (6)
Insomnia (Psychiatric disorders) | 15 (18) | 18 (23)
Dysuria (Renal and urinary disorders) | 9 (14) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (36) | 18 (27)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 13 (17)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 13 (20)
Alopecia (Skin and subcutaneous tissue disorders) | 38 (40) | 40 (50)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (10) | 6 (7)
Nail disorder (Skin and subcutaneous tissue disorders) | 9 (13) | 5 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 20 (42) | 14 (19)
Rash (Skin and subcutaneous tissue disorders) | 23 (35) | 12 (17)
Hot flush (Vascular disorders) | 9 (14) | 9 (17)
Hypertension (Vascular disorders) | 22 (54) | 24 (65)
Lymphoedema (Vascular disorders) | 7 (10) | 5 (5)
Haemorrhoids (Gastrointestinal disorders) | 7 (7) | 2 (2)
Paronychia (Infections and infestations) | 7 (12) | 3 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (17) | 5 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.